CLINICAL TRIAL: NCT04277377
Title: Donor-specific Anti-human Leukocyte Antigen Antibodies (DSA) Re-moval From Patient Blood Using Functionalized Nanoparticles - an ex Vivo Feasibility and Proof of Principle Study
Brief Title: Nanoparticle for DSA Removal
Status: Active, not recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00295
Record Dates: First submitted 2020-02-13; First posted 2020-02-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Kidney Failure; Presence of Donor Specific Antibodies
Keywords: Donor specific antibodies; Kidney transplantation; Coated nanoparticles
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bloodsample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- DSA in patients with kidney failure: Patients on kidney transplantation waiting list with DSA detected by Luminex (and mean fluorescence intensity (MFI) > 1000) in their blood.

SUMMARY:
Magnetic nanoparticles, coated with human leukocyte antigens (HLA) to capture anti-HLA antibodies with donor specificity (donor-specific antibodies, DSA), will be tested ex-vivo.

DETAILED DESCRIPTION:
This project aims at developing a new method using human leukocyte antigens (HLA)-coated magnetic nanoparticles to remove donor-specific antibodies (DSA) from the patients' blood ex vivo, while trying to keep the blood unaffected after exposure to the particles.

Nanoparticles will be engineered and tested ex vivo. While nanoparticles were successfully coated with macromolecules such as antibodies in the past, this is a new approach, which will be performed by the research group.

The goal of this project is to capture DSA in patient blood ex vivo and to remove them by magnetic separation. Efficacy and safety of this procedure will be assessed, especially the interaction of these novel particles with other blood components such as coagulation factors or effector cells, which could produce inflammatory mediators. According analyses are initiated and carried out.

ELIGIBILITY:
Inclusion Criteria:

* DSA in the blood as detected by Luminex®
* Adults (>18 years old)
* Informed written consent

Exclusion Criteria:

* Inability to follow the procedures of the study, due to language problems, psychological disorders, social conditions or dementia
* Pregnancy and/or breast feeding
* Unwillingness to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from kidney failure with DSA.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of DSA removed in a blood sample using HLA-coated magnetic nanoparticles | 1 day
  Quantification of DSA removal using HLA-coated magnetic nanoparticles in comparison with blood treated with control nanoparticles (without HLA coating).

SECONDARY OUTCOMES:
Blood coagulation (rotational thromboelastometry ROTEM, plasma clotting time) before and after treatment with HLA-coated magnetic nanoparticles | 1 day
  Coagulation parameters as described will be evaluated in blood samples. The same analyses will be repeated after exposure to HLA-coated magnetic nanoparticles.
Inflammatory blood mediators (IL-6, MCP-1) before and after treatment with HLA-coated magnetic nanoparticles | 1 day
  Inflammatory parameters as described will be evaluated in blood samples. The same analyses will be repeated after exposure to HLA-coated magnetic nanoparticles.

CONTACTS AND LOCATIONS:
Overall Officials: Beatrice Beck Schimmer, Prof, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Division of Anaesthesiology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wan SS, Ying TD, Wyburn K, Roberts DM, Wyld M, Chadban SJ. The Treatment of Antibody-Mediated Rejection in Kidney Transplantation: An Updated Systematic Review and Meta-Analysis. Transplantation. 2018 Apr;102(4):557-568. doi: 10.1097/TP.0000000000002049. PMID 29315141
- [Background] Herrmann IK, Beck-Schimmer B, Schumacher CM, Gschwind S, Kaech A, Ziegler U, Clavien PA, Gunther D, Stark WJ, Graf R, Schlegel AA. In vivo risk evaluation of carbon-coated iron carbide nanoparticles based on short- and long-term exposure scenarios. Nanomedicine (Lond). 2016 Apr;11(7):783-96. doi: 10.2217/nnm.16.22. Epub 2016 Mar 16. PMID 26979124
- [Background] Jacobson M, Roth Z'graggen B, Graber SM, Schumacher CM, Stark WJ, Dumrese C, Mateos JM, Aemisegger C, Ziegler U, Urner M, Herrmann IK, Beck-Schimmer B. Uptake of ferromagnetic carbon-encapsulated metal nanoparticles in endothelial cells: influence of shear stress and endothelial activation. Nanomedicine (Lond). 2015;10(24):3537-46. doi: 10.2217/nnm.15.172. Epub 2015 Oct 5. PMID 26434758